CLINICAL TRIAL: NCT06065605
Title: Pilot Study to Assess Clinical and Pivotal Biomarkers in the Urine to Predict the Progression of Nephropathy in Fabry Disease
Brief Title: Assess Urine Biomarkers to Predict Nephropathy in Fabry Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 23-LDRTC-01
Record Dates: First submitted 2023-09-11; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Fabry Disease
Keywords: Urine collection; biomarkers; CKD; Early detection
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Fabry patients without clinical evidence of nephropathy: No deterioration of kidney function.
- Fabry patients with clinical evidence of nephropathy: Deterioration of kidney function.
- Naïve Fabry patients: These patients have no received treatment.
- Healthy controls: Not diagnosed with Fabry disease.

SUMMARY:
The purpose of this research is to collect biological samples (urine) to develop assays for immune biomarkers to possibly in the future be able to screen subjects with Fabry disease and be able to understand better progression of nephropathy in Fabry disease and predict nephropathy in Fabry disease.

DETAILED DESCRIPTION:
This is a study to assess the markers related to autophagy, apoptosis, pyroptosis, and inflammatory markers related to NFkB, TNF-alpha, and TGF-β1 pathways in the urine. Urinary biomarkers will then be compared to the standard measures of kidney function and proteinuria: GFR, cystatin-C, B2M, bikunin, NGAL. Gb3 and Lyso-Gb3, urine microalbumin, and urine protein-to-creatinine (UPCR) ratio. Investigators will also analyze the role of therapy, especially for the inflammatory responses in participants on stable enzyme replacement therapy (ERT) with that of patients naïve to therapy.

There will be a total of 25 biomarkers that will be assessed during the study. Biomarkers of inflammation

1. Il-4
2. Il-6
3. IL-8
4. Il-10
5. Il-12
6. Il-18
7. MCP1
8. TGF-β1
9. IFN-γ
10. TNF-α
11. IL-1β
12. RANTES
13. BAFF
14. APRIL
15. PAI-1 Biomarkers of kidney function and proteinuria
16. B2M
17. Bikunin
18. NGAL
19. Osteopontin
20. Clusterin
21. Creatinine Acute kidney injury
22. KIM-1
23. YKL-40
24. EGF
25. CK-18 M30

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subject is greater than 18 but not older than 80 years.
* Subject willing to sign the informed consent and/or assent.
* Confirmed diagnosis of Fabry disease based on deficient α-Gal A enzymatic activity and molecular analysis demonstrating pathogenic variants in the GLA gene.

Exclusion Criteria:

* Any other known genetic condition associated with CKD.
* Evidence of hepatitis B or C infections or other chronic infectious diseases,
* Pregnancy or breastfeeding.
* Any other chronic condition, as per PI's discretion, that makes the subject ineligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There is no particular study population being investigated. Only patient with Fabry disease and healthy controls from across the world will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
identify urinary inflammatory biomarkers associated with nephropathy in Fabry disease, Units pg/ml | through study completion, an average of 2 years
  IL-1β, TNF-α, IL-6, Il-4, IL-8, Il-10, Il-12, Il-18, MCP1, RANTES, BAFF, APRIL, TGF-β1, INF-gamma, and PAI-1will be measured in urine.

SECONDARY OUTCOMES:
Identify biomarkers of renal glomerular function, tubular injury and endothelial dysfunction. Units pg/ml | through study completion, an average of 2 years
  B2M, GFR, albumin, cystatin C, osteopontin, clusterin, creatinine, EGF, NGAL, KIM-1, alpha-1-microglobulin, bikunin, YKL-40, CK-18 M30.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lysosomal & Rare Disorders Research & Treatment Center, Rockville, Maryland
  - Lysosomal & Rare Disorders Research & Treatment Center, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT06065605/Prot_000.pdf
  • Informed Consent Form (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT06065605/ICF_001.pdf